CLINICAL TRIAL: NCT03610607
Title: Shifting the Ratio of S. Cristatus vs. P. Gingivalis in Periodontitis Patients by Intense Education of Periodontal Health Maintenance
Brief Title: Intense Education of Periodontal Health Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meharry Medical College (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MeXie2018
Record Dates: First submitted 2018-07-17; First posted 2018-08-01 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Chronical Periodontitis, Ratio of P. Gingivalis and S. Cristatus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intense education of periodontal health maintenance (Active Comparator)
  Interventions: Behavioral: Intense education
- No intense education of periodontal health maintenance (Placebo Comparator)
  Interventions: Behavioral: Intense education

INTERVENTIONS:
Behavioral: Intense education — we will inform patients with their own data including the number of P. gingivalis and ratio of S. cristatus and P. gingivalis detected immediately after periodontal treatment and 3 month after the treatment. Explaining these data in detail, in terms that the patient can understand, are equally as important as teaching the plaque control techniques.

SUMMARY:
Investigators hypothesize that good oral hygiene may inhibit P. gingivalis, a keystone periodontal pathogen, entering mature dental plaque, which leads to a higher ratio of S. cristatus and P. gingivalis. Investigators will educate and train periodontitis patients following periodontal therapy to maintain periodontal health. Initial and intense education of periodontal health maintenance will be provided and the ratio of S. cristatus and P. gingivalis in dental plaques will be compared and analyzed for correlation between patient's execution of periodontal health maintenance and education tools or the ratio of S. cristatus and P. gingivalis.

DETAILED DESCRIPTION:
The periodontal health maintenance will be evaluated by plaque index, periodontal pocket, and gingival inflammation status. Participants will be assigned into two groups after the second dentist visit based on their execution of periodontal health maintenance. Participants whose number of P. gingivalis is unchanged or higher compared to that found at baseline will be considered poor maintenance. Those not having maintained a good dental hygiene will further be randomly assigned to two groups. One group will be given more intense oral health education, while the other one will receive the same education as post therapy. The result of intensive education and a shift in ratio of S. cristatus and P. gingivalis will then be measured for both groups at the third dentist visit (9 months after initial periodontal treatment) and the effectiveness of the intervention will be tested at this stage.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have > 16 teeth, 2 or more interproximal sites with CAL >4 mm and 2 or more with pocket depth >5 mm.

Exclusion Criteria:

* No scaling and root planing within the previous year or periodontal surgeries in the previous five years.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Improvement of periodontal condition | 9 month
  1. Improvement of periodontal condition Response to periodontal treatment will be determined by a composite measure including 1) Plaque Index; 2) Gingival index; 3) Cemento-enamel junction, gingival margin, probing, and bleeding on probing from six sites on all teeth. The patients will be considered to have improved, non-changed, and worsening periodontitis, according to clinical measurements and comparison them with those before treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participants data for all primary and secondary outcome measures will be made available.